CLINICAL TRIAL: NCT05354830
Title: The Effect of Foot Massage on Pain, Sleep Quality and Early Discharge in Patients Undergoing Spinal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Collaborators: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Eda Polat, Principle Investigator, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IstanbulMU15
Record Dates: First submitted 2022-04-17; First posted 2022-04-29 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Spinal Fusion; Pain, Postoperative
Keywords: Foot massage; Sleep quality; Spinal surgery; Postoperative pain
MeSH Terms: conditions — Pain, Postoperative; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Randomized controlled parallel groups
Who Masked: Investigator
Masking Description: It was planned as an open-label, blinded, randomized and controlled experimental study. A computer-assisted simple randomization method was used to distribute the groups homogeneously. For this purpose, 72 sets were created by using the functions available at the "https://www.random.org/integer-sets" internet address, and each of these sets included 8 participants, 4 participants from each study group. As the next operation, 72 sets were shown with 1 number each, and 9 numbers between 1 and 72 were generated using the "RANDOMLY SEARCH" function in Excel, and 9 sets to be used in randomization were randomly determined. In order to reach the sample number of 68 people, 4 participants, 2 from each study group, were selected in the final set. Thus, patients were randomly assigned to the experimental and control groups in order to reduce selection bias and control the variables that may affect the outcome parameters.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Foot Massage (Experimental): Patients undergoing TPF surgery and foot massage
  Interventions: Other: Foot Massage
- Control (No Intervention): Those who underwent TPF surgery and did not receive foot massage

INTERVENTIONS:
Other: Foot Massage — Foot Massage
  Arms: Foot Massage

SUMMARY:
In recent years, it is known that the use of complementary approaches, which are accepted as a safe and effective method for maintaining health and well-being, providing relaxation/relaxation, and reducing the effects of illness, has been increasing. It is reported that massage, which originates from an instinctive need for touch and is one of the oldest treatment methods, was first described in China in the second century BC and immediately after in India and Egypt, and was widely used by other early cultures such as Arabs, Greeks, Italians and Romans. In papyruses, on rocks, and in ancient oral stories dating back 15,000 years, there is evidence of the use of hands to provide comfort and healing. It is stated that foot massage, which is one of the most frequently used massage types today, has been applied in different parts of the world such as Egypt, India and China for thousands of years. In addition to pharmacological methods, non-pharmacological complementary and alternative treatment methods are also used in the control of pain due to reasons such as dissatisfaction with traditional treatment methods, reluctance to use invasive procedures and daily analgesics, and the toxic effects of drugs. Massage provides relaxation both physically and mentally. It is thought to reduce edema by accelerating circulation, muscle tension and anxiety by the stimuli reaching the spinal cord, and pain sensation by stimulating peripheral sensory receptors.

DETAILED DESCRIPTION:
In recent years, it is known that the use of complementary approaches, which are accepted as a safe and effective method for maintaining health and well-being, providing relaxation/relaxation, and reducing the effects of illness, has been increasing. It is reported that massage, which originates from an instinctive need for touch and is one of the oldest treatment methods, was first described in China in the second century BC and immediately after in India and Egypt, and was widely used by other early cultures such as Arabs, Greeks, Italians and Romans. In papyruses, on rocks, and in ancient oral stories dating back 15,000 years, there is evidence of the use of hands to provide comfort and healing. It is stated that foot massage, which is one of the most commonly used types of massage today, has been applied in different parts of the world such as Egypt, India and China for thousands of years. It is stated that Ibn-i Sina talked about the benefits of massage and included this subject in the world-famous source of information, El Kanun Fi't Medicine. It is reported that massage therapy started to be applied in the USA in the mid-1800s and continued its development by using it for different purposes, while in England, nine nurses came together and founded the Massage Association in 1894. In Turkey, it is stated that massage was first applied in Gülhane Serriyat Hospital in 1909 by physical therapists for treatment purposes. Spinal stabilization and fusion techniques for various pathological conditions of the spine began in the 1990s and have now become a surgical standard. The main purpose of surgical treatment in spinal disorders; to correct spinal deformity, increase spinal fusion rates, provide neurological decompression, ensure normal stability, and facilitate rehabilitation by reducing pain following surgery. He has defined many surgical intervention methods for the spine, and these are roughly classified as anterior, posterior and lateral intervention methods. Among these methods, posterior intervention methods are used most frequently. Posterior spine stabilization; It is performed using transpedicular screw and posterior bone fusion. Surgical intervention in degenerative disc disease; It can be applied with open and percutaneous fixation techniques. Transpedicular fixation (TPF); It is one of the most effective surgical methods in the treatment of spinal instability in terms of providing anatomical reduction, stable fixation and early mobilization. It immobilizes the mobile segment of the spine by allowing adequate decompression of neural structures and ensuring bone fusion. Screws in transpedicular fixation surgery; It can be implanted at different levels of the spine such as the cervical, thoracic, lumbar and sacral regions. Pain is a part of the common experiences that people live most of the time, and it is a complex sensation that affects people, is affected by individual characteristics, is always subjective, subjective, and difficult to understand and define. Pain affects the life of the individual physically, mentally and socially and reduces the quality of life of individuals. Therefore, controlling the pain experienced by individuals is important in terms of relaxation of the individual, increasing the quality of life, reducing complications and shortening the length of hospital stay. Today, pharmacological methods are widely used in the control of pain. However, when analgesics are used unconsciously and intensively, they have a negative effect on some physiological functions; Especially in cases where narcotics are used, undesirable situations such as tolerance development due to increasing the dose are encountered each time. In addition to pharmacological methods, non-pharmacological complementary and alternative treatment methods are also used in the control of pain due to reasons such as dissatisfaction with traditional treatment methods, reluctance to use invasive procedures and daily analgesics, and the toxic effects of drugs. Massage provides relaxation both physically and mentally. It is thought that it reduces edema by accelerating circulation, muscle tension and anxiety when stimuli reach the spinal cord, and pain sensation by stimulating peripheral sensory receptors. As with every surgical procedure, intense postoperative pain occurs especially after spinal surgery. Many factors play a role in the emergence of this pain. One of these is the postoperative inflammatory tissue response. Another factor is the long-term use of automatic retractor systems placed on the paravertebral muscles during spinal surgery. Undesirable severe low back pain in the postoperative period due to prolonged paravertebral muscle retraction is a common and distressing condition for both the patient and the surgeon in the early postoperative period. Therefore, intensive and strong analgesic treatments and even narcotic analgesics have to be used in the early postoperative period. It is stated that pain increases the level of depression, this situation lowers the pain threshold and negatively affects sleep quality in pain and depression. Sleep disorders reduce the quality of life; It increases the risk of falling, the cost of treatment, and most importantly, the death rate in patients. Foot massage provides the transfer of sensory stimuli to the brain by stimulating the nervous system and increasing dopamine secretion. The advantages of foot massage are that it is easy to apply, inexpensive, and no special equipment is needed. Studies on pain and anxiety management with foot massage; shows that it is possible to reduce the pain of patients with this method.

ELIGIBILITY:
Inclusion Criteria:

* Having TPF surgery,
* Be over 18 years old,
* No nerve damage or psychiatric disease in the history,
* No central nervous system metastasis or disease,
* No irritation or ulceration in the skin area to be massaged,
* No history of deep vein thrombosis
* To be able to speak and understand Turkish and to be able to read and write,
* Patients with an ASA score of 1 and 2,
* It is voluntary to participate in the research.

Exclusion Criteria:

* Not wanting to leave the study for any reason,
* Patients with an ASA score of 3 and above,
* Complication development.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Pain Visual Analogue Scale | 12 months
  The highest score that can be obtained from the visual analog scale is 10 and the lowest 0. As the higher score is obtained, the patient's pain will increase, and the result is evaluated as bad.
  Visual Analogue Scale scores will decrease after progressive muscle relaxation exercises. The highest score that can be obtained from the visual analog scale is 10 and the lowest 0. As the higher score is obtained, the patient's pain will increase, and the result is evaluated as bad.
  Visual Analogue Scale scores will decrease after progressive muscle relaxation exercises. The highest score that can be obtained from the visual analog scale is 10 and the lowest 0. As the higher score is obtained, the patient's pain will increase, and the result is evaluated as bad.
Sleep Richard-Campbell Sleep Questionnaire | 12 months
  A score of "0-25" from the scale indicates that the scale is very bad, and a score of "76-100" indicates that the scale is very good.

CONTACTS AND LOCATIONS:
Locations (1):
- Sultan 2. Abdülhamid Han Training and Research Hospital, Istanbul, Üsküdar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The work will not be shared after publication.

REFERENCES:
- [Background] Abbaspoor Z, Akbari M, Najar S. Effect of foot and hand massage in post-cesarean section pain control: a randomized control trial. Pain Manag Nurs. 2014 Mar;15(1):132-6. doi: 10.1016/j.pmn.2012.07.008. Epub 2013 Jan 24. PMID 23352729
- [Background] Ali ZS, Ma TS, Ozturk AK, Malhotra NR, Schuster JM, Marcotte PJ, Grady MS, Welch WC. Pre-optimization of spinal surgery patients: Development of a neurosurgical enhanced recovery after surgery (ERAS) protocol. Clin Neurol Neurosurg. 2018 Jan;164:142-153. doi: 10.1016/j.clineuro.2017.12.003. Epub 2017 Dec 8. PMID 29232645
- [Background] Bagheri-Nesami M, Shorofi SA, Zargar N, Sohrabi M, Gholipour-Baradari A, Khalilian A. The effects of foot reflexology massage on anxiety in patients following coronary artery bypass graft surgery: a randomized controlled trial. Complement Ther Clin Pract. 2014 Feb;20(1):42-7. doi: 10.1016/j.ctcp.2013.10.006. Epub 2013 Oct 25. PMID 24439644
- [Background] Cuschieri RJ, Morran CG, Howie JC, McArdle CS. Postoperative pain and pulmonary complications: comparison of three analgesic regimens. Br J Surg. 1985 Jun;72(6):495-8. doi: 10.1002/bjs.1800720631. PMID 4016522
- [Background] Deyo RA, Mirza SK, Martin BI, Kreuter W, Goodman DC, Jarvik JG. Trends, major medical complications, and charges associated with surgery for lumbar spinal stenosis in older adults. JAMA. 2010 Apr 7;303(13):1259-65. doi: 10.1001/jama.2010.338. PMID 20371784
- [Background] Emslie MJ, Campbell MK, Walker KA. Changes in public awareness of, attitudes to, and use of complementary therapy in North East Scotland: surveys in 1993 and 1999. Complement Ther Med. 2002 Sep;10(3):148-53. doi: 10.1016/s0965229902000663. PMID 12568143
- [Background] Grealish L, Lomasney A, Whiteman B. Foot massage. A nursing intervention to modify the distressing symptoms of pain and nausea in patients hospitalized with cancer. Cancer Nurs. 2000 Jun;23(3):237-43. doi: 10.1097/00002820-200006000-00012. PMID 10851775
- [Background] Eadie J, van de Water AT, Lonsdale C, Tully MA, van Mechelen W, Boreham CA, Daly L, McDonough SM, Hurley DA. Physiotherapy for sleep disturbance in people with chronic low back pain: results of a feasibility randomized controlled trial. Arch Phys Med Rehabil. 2013 Nov;94(11):2083-92. doi: 10.1016/j.apmr.2013.04.017. Epub 2013 May 2. PMID 23643716
- [Background] Lu WA, Chen GY, Kuo CD. Foot reflexology can increase vagal modulation, decrease sympathetic modulation, and lower blood pressure in healthy subjects and patients with coronary artery disease. Altern Ther Health Med. 2011 Jul-Aug;17(4):8-14. PMID 22314629
- [Background] Mahdavipour F, Rahemi Z, Sadat Z, Ajorpaz NM. The effects of foot reflexology on depression during menopause: A randomized controlled clinical trial. Complement Ther Med. 2019 Dec;47:102195. doi: 10.1016/j.ctim.2019.102195. Epub 2019 Sep 14. PMID 31780002